CLINICAL TRIAL: NCT07128628
Title: A 4-Week, Randomized, Double-Masked, Parallel-Group, Active-Controlled, Multicenter Study Evaluating Lifitegrast/Perfluorohexyloctane Fixed-Dose Combination Administered Twice Daily on Signs and Symptoms of Dry Eye Disease
Brief Title: A Study Evaluating the Safety and Efficacy of a Fixed-Dose Combination for Dry Eye Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BL-RX01-OPUSNG-1201
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast; perfluorohexyl-octan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Experimental)
  Interventions: Drug: Lifitegrast/Perfluorohexyloctane Fixed Dose Combination
- Arm 2 (Active Comparator)
  Interventions: Drug: Lifitegrast
- Arm 3 (Active Comparator)
  Interventions: Drug: Perfluorohexyloctane
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Vehicle
- Arm 5 (Placebo Comparator)
  Interventions: Drug: Vehicle
- Arm 6 (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Lifitegrast/Perfluorohexyloctane Fixed Dose Combination — Topical ocular drop of lifitegrast and perfluorohexyloctane administered for 4 weeks
  Arms: Arm 1
Drug: Lifitegrast — Topical ocular drop of lifitegrast administered for 4 weeks
  Arms: Arm 2
Drug: Perfluorohexyloctane — Topical ocular drop of perfluorohexyloctane administered for 4 weeks
  Arms: Arm 3
Drug: Vehicle — Topical ocular drop with no active ingredients administered for 4 weeks
  Arms: Arm 4
Drug: Vehicle — Topical ocular drop with no active ingredients administered for 4 weeks
  Arms: Arm 5
Drug: Vehicle — Topical ocular drop with no active ingredients administered for 4 weeks
  Arms: Arm 6

SUMMARY:
A 4-Week, Randomized, Double-Masked, Parallel-Group, Active-Controlled, Multicenter Study Evaluating Lifitegrast/Perfluorohexyloctane Fixed-Dose Combination Administered Twice Daily on Signs and Symptoms of Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

This study will include subjects who meet all of the following inclusion criteria:

* Voluntarily provide written informed consent
* ≥18 years of age
* Subject-reported history of DED OU for at least 6 months
* Same eye satisfies the following criteria for dry eye signs at both screening and baseline/randomization
* The criteria for dry eye symptoms are met at both screening and baseline/randomization
* As needed (PRN) or scheduled use of non-prescription (OTC) artificial tear, gels, or lubricants for symptoms of dry eye within the past 30 days
* Able and willing to follow instructions, including participation in all trial assessments and visits

Exclusion Criteria:

This study will exclude subjects who meet any of the following exclusion criteria (Note: Ocular exclusion criteria are relevant to both eyes, such that meeting a criterion in either eye excludes the subject from the study):

* Known allergy or sensitivity to any study treatment (or any of its components)
* Best-corrected visual acuity (BCVA) of 0.7 logarithm of the minimum angle of resolution (logMAR) or worse (50 Early Treatment Diabetic Retinopathy Study [ETDRS] letters; Snellen equivalent score of 20/100 or worse) at Visit 1 (Screening) or Visit 2 (baseline/randomization)
* Any clinically significant (CS) ocular surface slit-lamp findings at Visit 1 (Screening) or Visit 2 (baseline/randomization), or findings that may interfere with trial parameters in the opinion of the Investigator.
* Use of any of any ocular therapies within 30 days.
* Unable or unwilling to stop current topical dry eye treatments

Additional criteria per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Total corneal fluorescein staining change from baseline | Baseline, day 29

IPD SHARING:
Plan to Share IPD: No